CLINICAL TRIAL: NCT05806892
Title: The Effect of Warm Application to the Breast With the Help of Thera Pearl in the Postpartum Period on Milk Release, Breastfeeding Success of Mothers, Milk Perception and Postpartum Breastfeeding Self-Efficacy: A Randomized Controlled Study
Brief Title: The Effect of Warm Application to the Breast With the Aid of Thera Pearl on Milk Release and Breastfeeding Success
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amasya University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AmasyaU-betuluzun-002
Record Dates: First submitted 2023-03-11; First posted 2023-04-10 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Breast Feeding
Keywords: postpartum period; Thera Pearl; Breastfeeding Self-Efficacy; randomized controlled trial
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: The first interview with women who gave birth will be held in the postpartum service of the relevant hospital. In this interview, Personal Information Form, Breastfeeding Observation Form (for the first 24 hours after birth), Bristol Breastfeeding Evaluation Scale, Breastfeeding Self-Efficacy Scale and Insufficient Milk Perception Scale will be filled. At the same time, the phone and address information of the participants will be obtained in this meeting, and the postpartum 2-7. and 10-15. You will be informed that there will be a home visit on days.
  Thera Pearl application will be explained to the woman in detail and the first application will be carried out together in the hospital.
  Then the participant is postpartum 2-7. on days and 10-15. They will be visited at home once a day and their status of applying Thera Pearl will be questioned. The final test will be applied.
Who Masked: Participant
Masking Description: It is aimed to blind the puerperant women participating in the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): Thera Pearl application will be explained to the woman in detail and the first application will be carried out together in the hospital.
  Interventions: Other: Thera Pearl
- Control (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Other: Thera Pearl — You can apply Thera°Pearl warm breast therapy before breastfeeding or during milking. You should do this application 4 times a day, in the morning, at noon, in the evening and at night before going to bed. Each application should be done on both breasts and should last at least 20 minutes.
  Thera°Pearl Warm Breast Therapy has been developed to open milk ducts and accelerate milk flow.
  Thermogel packs for Thera°Pearl hot therapy can be heated inside the fabric covers in the microwave for a maximum of 15 seconds or in hot water by removing the fabric covers. Packages that have been removed from the cover should be kept in boiling water for 1-2 minutes and then applied by putting them into the sheath.
  Arms: Experiment

SUMMARY:
Breastfeeding and breast milk are very important in supporting newborn growth and development. The World Health Organization (WHO) and the United Nations Children's Fund (UNICEF) recommend that breastfeeding should be continued with only breast milk for the first 6 months after birth and with complementary foods until the age of 2 years. However, the rate of breastfeeding all over the world is far from the targeted values. For this reason, it is necessary to plan and implement various interventions in order to start breastfeeding in the early period and to help maintain breastfeeding.

There are various problems associated with breastfeeding. Large, sunken or flat nipples, tongue-tie in the fetus, excessive milk production, lack of milk production or late onset are some of these problems. It is known that the most common problems are breast fullness or late onset of milk production. In both cases, early resolution is important in ensuring the sustainability of breastfeeding. During the breastfeeding period, various applications are used in order to both relieve fullness and increase milk production. Applying hot water to the udder is the most preferred way to increase milk production. The fact that it does not require much cost, does not contain any herbal or pharmacological agents and is easy to apply, as well as relieving the fullness of the breasts for the mother and increasing milk production, increases the popularity of hot water application. When the relevant literature was reviewed, it was seen that the hot application to the breast was generally done through a warm towel or hot water bag, but there was no study using Thera Pearl.

This study will be carried out in an experimental design in order to evaluate the effect of warm application applied to the breast with the help of Thera Pearl in the postpartum period on milk release, breastfeeding success of mothers, milk perception and postpartum breastfeeding self-efficacy. The research will be carried out in Amasya University Sabuncuoğlu Şerefeddin Training and Research Hospital obstetrics service between April and September 2023. Personal Information Form, Breastfeeding Observation Form, Bristol Breastfeeding Evaluation Scale, Breastfeeding Self-Efficacy Scale and Insufficient Milk Perception Scale will be used to collect data. It is thought that the application to be made for breastfeeding problems and milk release will be effective.

DETAILED DESCRIPTION:
Breastfeeding and breast milk are very important in the protection and development of maternal and newborn health. Breast milk is a nutrient with unique immunological and anti-inflammatory properties that protect against many diseases. The World Health Organization and the United Nations Children's Fund recommend continuing breastfeeding with appropriate complementary foods until the age of 2, without any additional food for the first six months after birth, as the first condition of a healthy diet.

The World Health Organization announced that the rate of exclusive breastfeeding in the first six months is 44% worldwide in 2020. UNICEF reported that one in five babies in high-income countries and one in 25 babies in low- and middle-income countries are not breastfed at all.

Breastfeeding problems may occur for various reasons in the postpartum period. Breast fullness or late onset of milk production are among the most common of these problems. In cases where milk production is too high, breast fullness can be experienced, while milk production can be very slow in the opposite case. In both cases, early resolution is important in ensuring the sustainability of breastfeeding. The absence or late onset of milk production after birth causes the mother to be alarmed, interruption of breastfeeding, and ultimately feeding the newborn with formula. In the first 6 months of life, when the baby should receive only breast milk, feeding with formulas other than breast milk or different nutrients is an issue that needs to be addressed as it will adversely affect its growth and development. In this sense, milk production should be supported by making use of non-pharmacological methods in the postpartum period. Massage, herbal agents or hot water application are often preferred to increase milk production. Applying hot water to the udder is the most preferred way to increase milk production. The fact that it does not require much cost, does not contain any herbal or pharmacological agents and is easy to apply, also relieves the fullness of the breasts for the mother and increases milk production, increases the popularity of hot water application. As a matter of fact, in a study, it was determined that women who applied hot water to the nipples in the first 10 days after giving birth experienced less pain. When the relevant literature was reviewed, it was seen that there was no study using Thera Pearl, in which the warm application to the breast was usually done through a warm towel or hot water bag.

For the experimental group:

The first interview with women who gave birth will be held in the postpartum service of the relevant hospital. In this interview, Personal Information Form, Breastfeeding Observation Form (for the first 24 hours after birth), Bristol Breastfeeding Evaluation Scale, Breastfeeding Self-Efficacy Scale and Insufficient Milk Perception Scale will be filled. At the same time, the phone and address information of the participants will be obtained in this meeting, and the postpartum 2-7. and 10-15. You will be informed that there will be a home visit on days.

Thera Pearl application will be explained to the woman in detail and the first application will be carried out together in the hospital.

Then the participant is postpartum 2-7. on days and 10-15. They will be visited at home once a day and their status of applying Thera Pearl will be questioned. In addition, the Breastfeeding Observation Form (for postpartum days 2-7 and 10-15), Bristol Breastfeeding Evaluation Scale, Breastfeeding Self-Efficacy Scale and Insufficient Milk Perception Scale will be filled again.

For the control group:

No intervention will be applied to the control group. The first interview with women who gave birth will be held in the postpartum service of the relevant hospital. In this interview, Personal Information Form, Breastfeeding Observation Form (for the first 24 hours after birth), Bristol Breastfeeding Evaluation Scale, Breastfeeding Self-Efficacy Scale and Insufficient Milk Perception Scale will be filled. At the same time, the phone and address information of the participants will be obtained in this meeting, and the postpartum 2-7. and 10-15. You will be informed that home visits will be made on the following days.

Then the participant is postpartum 2-7. and 10-15. Breastfeeding Observation Form (for postpartum days 2-7 and 10-15), Bristol Breastfeeding Evaluation Scale, Breastfeeding Self-Efficacy Scale and Insufficient Milk Perception Scale will be filled in once a day.

ELIGIBILITY:
Inclusion Criteria:

* Being a primary school graduate
* be over 18 years old
* Living in the city center of Amasya
* Being primiparous
* Being open to communication
* Those who volunteered to participate in the research
* Those with normal mental health

Exclusion Criteria:

* not willing to participate in research
* have any disease
* those who are not with the baby

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-07-24 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Bristol Breastfeeding Assessment Tool (BBAT): | within 24 hours of postpartum
  BBAT: The scale consists of 4 items. Each item is scored between 0-2 points. For each item, 0 points/poor, 1 point/moderate, 2 points/good are evaluated. The lowest score obtained from the scale is 0, and the highest score is 8. Low scores indicate that breastfeeding is not effective, while high scores indicate that breastfeeding is effective.
Breast-feeding Self-efficacy Scale (BSS) | within 24 hours of postpartum
  BSS: The minimum score that can be obtained from the scale is 14, and the maximum score is 70. The higher the score, the higher the breastfeeding self-efficacy.
Poor Milk Perception Scale (PMPS): | within 24 hours of postpartum
  PMPS: A minimum of 0 and a maximum of 50 points can be obtained from the scale. The higher the total score obtained, the higher the perception of milk adequacy.
Evaluation of Thera Pearl application 1 | within 2-7 days postpartum
  Bristol Breastfeeding Assessment Tool (BBAT): The scale consists of 4 items. Each item is scored between 0-2 points. For each item, 0 points/poor, 1 point/moderate, 2 points/good are evaluated. The lowest score obtained from the scale is 0, and the highest score is 8. Low scores indicate that breastfeeding is not effective, while high scores indicate that breastfeeding is effective.
Evaluation of Thera Pearl application 2 | within 2-7 days postpartum
  Breast-feeding Self-efficacy Scale (BSS): The minimum score that can be obtained from the scale is 14, and the maximum score is 70. The higher the score, the higher the breastfeeding self-efficacy.
Evaluation of Thera Pearl application 3 | within 2-7 days postpartum
  Poor Milk Perception Scale (PMPS): A minimum of 0 and a maximum of 50 points can be obtained from the scale. The higher the total score obtained, the higher the perception of milk adequacy.
Evaluation of Thera Pearl application 1 | within 10-15 days postpartum
  Bristol Breastfeeding Assessment Tool (BBAT): The scale consists of 4 items. Each item is scored between 0-2 points. For each item, 0 points/poor, 1 point/moderate, 2 points/good are evaluated. The lowest score obtained from the scale is 0, and the highest score is 8. Low scores indicate that breastfeeding is not effective, while high scores indicate that breastfeeding is effective.
Evaluation of Thera Pearl application 2 | within 10-15 days postpartum
  Breast-feeding Self-efficacy Scale (BSS): The minimum score that can be obtained from the scale is 14, and the maximum score is 70. The higher the score, the higher the breastfeeding self-efficacy.
Evaluation of Thera Pearl application 3 | within 10-15 days postpartum
  Poor Milk Perception Scale (PMPS): A minimum of 0 and a maximum of 50 points can be obtained from the scale. The higher the total score obtained, the higher the perception of milk adequacy.

CONTACTS AND LOCATIONS:
Overall Officials: Hava Özkan, Özkan, Principal Investigator — Ataturk University

IPD SHARING:
Plan to Share IPD: Yes
It is planned to publish the obtained data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: It is planned that the data obtained will be published within 4 months.
Access Criteria: The article published in a journal suitable for the research topic can be read by the members of the journal.